CLINICAL TRIAL: NCT02041286
Title: User Performance of the Karajishi Contour Blood Glucose Monitoring System
Brief Title: Evaluation of an Karajishi Contour Investigational Blood Glucose Monitoring System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ascensia Diabetes Care (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: GCA-2013-001-01
Record Dates: First submitted 2014-01-17; First posted 2014-01-22 (Estimated); Results first posted 2015-06-19 (Estimated); Last update posted 2016-02-29 (Estimated); Status verified 2016-01

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intended Users of the Monitoring System (Experimental): Subjects with diabetes use the Karajishi Contour Investigational BG Monitoring System with no training. The criteria for the intended use population:
  1. At least 60% of subjects will be younger than age 65
  2. At least 10% of subjects will have type 1 diabetes
  Interventions: Device: Karajishi Contour Investigational BG Monitoring System

INTERVENTIONS:
Device: Karajishi Contour Investigational BG Monitoring System — Subjects with diabetes perform self Blood Glucose (BG) tests with capillary fingerstick and palm blood using the Karajishi Contour Investigational BG Monitoring System with no training. All BG results are compared to reference method results obtained from subject capillary plasma. Also, study staff test subject venous blood and BG results are compared to reference method results obtained from subject venous plasma.

SUMMARY:
The purpose of this study is to determine if subjects who have diabetes can operate the Investigational Blood Glucose Monitoring System (BGMS) without training and obtain valid glucose results.

ELIGIBILITY:
Inclusion Criteria:

* Males and females, 18 years of age and older
* People with type 1 or type 2 diabetes
* Able to speak, read, and understand English
* Willing to complete all study procedures

Exclusion Criteria:

* Hemophilia or any other bleeding disorder
* Pregnancy
* Physical, visual, or neurological impairments that would make the person unable to perform testing with the BGM
* Previously participated in a BG monitor study using the Karajishi BGMS (or used a Bayer Contour meter)
* Working for a medical laboratory, hospital, or other clinical setting that involves training on and clinical use of blood glucose monitors
* Working for a competitive medical device company, or having an immediate family member who works for such a company
* A condition which, in the opinion of the investigator or designee, would put the person or study conduct at risk

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2014-01; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leslie J Klaff, MD, Principal Investigator — Rainier Clinical Research Center; Timothy Bailey, MD, Principal Investigator — AMCR Institute
Locations (2):
- United States (2):
  - AMCR Institute, Escondido, California
  - Rainier Clinical Research Center, Renton, Washington

RESULTS

PARTICIPANT FLOW:
Groups:
- Intended Users of the Monitoring System: Subjects with diabetes use the Karajishi Contour Investigational BG Monitoring System with no training. The criteria for the intended use population:
  1. At least 60% of subjects will be younger than age 65
  2. At least 10% of subjects will have type 1 diabetes
  Karajishi Contour Investigational BG Monitoring System: Subjects with diabetes perform self Blood Glucose (BG) tests with capillary fingerstick and palm blood using the Karajishi Contour Investigational BG Monitoring System with no training. All BG results are compared to reference method results obtained from subject capillary plasma. Also, study staff test subject venous blood and BG results are compared to reference method results obtained from subject venous plasma.
Period: Overall Study
Arm/Group | Intended Users of the Monitoring System
Started | 136
Completed | 135 (One subject discontinued from testing after low BG fingerstick result (hypoglycemia AE).)
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Groups:
- Intended Users of the Monitoring System: Subjects with diabetes use the Karajishi Contour Investigational BG Monitoring System with no training.
Arm/Group | Intended Users of the Monitoring System
Number analyzed (Participants) | 136
Age, Customized [Mean (Full Range); unit: years]
  Age of enrolled subjects | 52.5 [18 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 63
  Male | 73
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 130
  Unknown or Not Reported | 1
Race (NIH/OMB) [Number; unit: participants] — Subjects provided more than one choice for Race, therefore the apparent frequency total for Race was different from number of subjects.
  participants
    American Indian or Alaska Native | 2
    Asian | 7
    Native Hawaiian or Other Pacific Islander | 1
    Black or African American | 10
    White | 118
    More than one race | 3
    Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 136

OUTCOME MEASURES:

1. Primary Outcome: Number of Self-Test Fingerstick Blood Glucose (BG) Results Within +/- 15 mg/dL (<100 mg/dL) and Within +/- 15% (>=100 mg/dL) of Laboratory Glucose Method
Description: Subjects with diabetes self-test fingerstick blood use an investigational Blood Glucose Monitoring System (BGMS) with no training. BGMS results are compared with subject capillary plasma BG results obtained with a Yellow Springs Instrument (YSI) Analyzer. YSI Analyzer BG results are used to calculate the number of BGMS results within +/-15 mg/dL (<100 mg/dL YSI capillary plasma) and +/-15% (>=100 mg/dL YSI capillary plasma).
Time Frame: 1 hour
Population: 135 (136-1) Blood glucose results were analyzed. One subject discontinued from testing after low BG fingerstick result (hypoglycemia AE), thus no reference result available.
Measure: Number; unit: Blood glucose results
Arm/Group | Intended Users of the Monitoring System
Number analyzed (Participants) | 135
Blood glucose results | 127

2. Secondary Outcome: Number of Venous Blood Glucose (BG) Results Within +/- 15 mg/dL (<100 mg/dL) and Within +/- 15% (>=100 mg/dL) of Laboratory Glucose Method
Description: Study staff test subject venous blood using an investigational Blood Glucose Monitoring System (BGMS). Venous BGMS results are compared with subject venous plasma BG results obtained with a Yellow Springs Instrument (YSI) Analyzer. YSI Analyzer venous plasma BG results are used to calculate the number of BGMS results within +/-15 mg/dL (<100 mg/dL YSI venous plasma) and +/-15% (>=100 mg/dL YSI venous plasma).
Time Frame: 1 hour
Population: 132 (136-4) Blood glucose results were analyzed. One subject discontinued from all testing after hypoglycemia AE. One (1) subject lab reference replicates were discrepant and not evaluable per protocol. Venipuncture was not successful for 2 subjects.
Measure: Number; unit: Blood glucose results
Groups:
- Intended Users of the Monitoring System: Study staff test subject venous blood and BG results are compared to reference method results obtained from subject venous plasma.
Arm/Group | Intended Users of the Monitoring System
Number analyzed (Participants) | 132
Blood glucose results | 131

3. Secondary Outcome: Number of Blood Glucose (BG) Results From Alternative Site Testing (AST) Palm Blood Within +/- 15 mg/dL (<100 mg/dL) and Within +/- 15% (>=100 mg/dL) of Laboratory Glucose Method
Description: Subjects with diabetes self-test Alternative Site (AST) palm blood using an investigational Blood Glucose Monitoring System (BGMS) with no training. BGMS AST palm results are compared with subject capillary plasma BG results obtained with a Yellow Springs Instrument (YSI) Analyzer. YSI Analyzer BG results are used to calculate the number of BGMS results within +/-15 mg/dL (<100 mg/dL YSI capillary plasma) and +/-15% (>=100 mg/dL YSI capillary plasma).
Time Frame: 1 hour
Population: 130 (136-6) Blood glucose results were analyzed. One subject discontinued from all testing after hypoglycemia AE. One (1) subject with low blood sugar did not attempt AST testing per protocol. No AST palm results were obtained for one (1) subject. Three (3) subjects had low blood sugar; AST results were not evaluable per protocol.
Measure: Number; unit: Blood glucose results
Arm/Group | Intended Users of the Monitoring System
Number analyzed (Participants) | 130
Blood glucose results | 112

4. Secondary Outcome: Number of Subject Fingerstick Blood Glucose (BG) Results Within +/- 15 mg/dL (<100 mg/dL) and Within +/- 15% (>=100 mg/dL) of Laboratory Glucose Method When Obtained and Tested by Study Staff
Description: Study staff obtain and test subject fingerstick blood using an investigational Blood Glucose Monitoring System (BGMS). BGMS results are compared with subject capillary plasma BG results obtained with a Yellow Springs Instrument (YSI) Analyzer. YSI capillary plasma results are used to calculate the number of BGMS results within +/-15 mg/dL (<100 mg/dL YSI capillary plasma) and +/-15% (>=100 mg/dL YSI capillary plasma).
Time Frame: 1 hour
Population: 135 (136-1) Blood glucose results were analyzed. One subject discontinued from all testing after hypoglycemia AE.
Measure: Number; unit: Blood glucose results
Groups:
- Intended Users of the Monitoring System: Study staff test subject capillary blood and BG results are compared to reference method results obtained from subject capillary plasma.
Arm/Group | Intended Users of the Monitoring System
Number analyzed (Participants) | 135
Blood glucose results | 133

5. Secondary Outcome: Number of Subject Responses That Strongly Agree or Agree or Are Neutral With Questionnaire Statements
Description: Staff will obtain subject responses using short questionnaires to provide feedback on instructions for use and the basic operation of the BGMS. Subjects may respond Strongly Agree; Agree; Neutral; Disagree; or Strongly Disagree.
Time Frame: 1 hour
Measure: Number; unit: participants
Arm/Group | Intended Users of the Monitoring System
Number analyzed (Participants) | 136
participants
  I find it easy to do a blood test with this meter. | 136
  The meter display is easy to see and read. | 136
  It is easy to understand my test results. | 136
  I like the overall meter design. | 136
  I find the meter easy to use. | 136
  The instruction (User Guide) is easy to understand | 136
  Instructions clearly explain how to run a test. | 136
  Instructions clearly explain meter error messages. | 136

ADVERSE EVENTS:
Time Frame: 1 hour subject visit
Arm/Group | Intended Users of the Monitoring System
Serious Adverse Events (participants affected / at risk) | 0/136
Other Adverse Events (participants affected / at risk) | 4/136
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intended Users of the Monitoring System (N=136)
Hypoglycemia (Endocrine disorders) | 4 (4) — One subject discontinued from all testing after hypoglycemia AE. Subject's hypoglycemia was resolved at the visit.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days